CLINICAL TRIAL: NCT01646801
Title: The Use of NMB Drug Ejecting Balloon for Treatment of Patients With Peripheral Arterial Disease
Brief Title: Study of NMB Drug Ejecting Balloon for Peripheral Arteries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: N.M.B. Medical Applications Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMB PP CLD 2158
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (1):
- Experimental (Experimental): NMB's Paclitaxel Drug ejecting balloon catheter
  Interventions: Device: NMB Balloon Catheter

INTERVENTIONS:
Device: NMB Balloon Catheter — patients treated by the NMB's Drug Ejecting Balloon

SUMMARY:
The purpose of this study is to demonstrate the Safety and effectiveness of the use of NMB's drug ejecting balloon for the treatment of de novo and restenotic lesions in peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patient with lifestyle limiting claudication or rest pain (Rutherford- Becker scale 2, 3 or 4).
* Patient with de novo lesion or restenotic lesion ≥70% in the iliac, femoral, popliteal or tibial artery.
* The target lesion can be successfully crossed with a guide wire and dilated.
* The target lesion is in a native artery of 2.5-10mm in diameter and less than 80 mm in length.
* Patient is willing to and able to sign a written informed consent and to comply with procedures (e.g., adherence to follow-up visits, including 6 months CT-angiography/MRA follow-up).

Exclusion Criteria:

* Women who are pregnant or breast-feeding and women of childbearing potential who do not use adequate contraception.
* Previous participation in another study with any investigational drug or device within the past 30 days.
* The patient is currently enrolled in another investigational device or drug trial.
* Severe reaction to contrast agents that cannot be adequately premedicated prior to procedure.
* Stenosis with corresponding thrombosis treated within 7 days before enrollment.
* Patient with known contraindications for aspirin or other anticoagulant/antiplatelet therapy.
* Patient that has co-morbid illness that may result in life expectancy of less than 12 months.
* History of haemorrhagic stroke or gastro-intestinal bleeding within 6 months.
* Patient with major surgery during the 30 days preceding the interventional procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) | 6 months
  Late Lumen Loss (LLL) defined as the difference between the minimal luminal diameter after the procedure and at 6 months, as evaluated by Quantitative Angiography (mm units will be used)

SECONDARY OUTCOMES:
Restenosis rate | 6 months
  Restenosis is defined as stenosis of at least 50% of the luminal diameter at 6 months
Device Malfunction | intraprocedural, 3, 6 and 12 months
Adverse events | intraprocedural, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Rabin Medical Center, Hasharon Hospital, Petah Tikva, Israel